CLINICAL TRIAL: NCT01951664
Title: Feasibility and Preliminary Efficacy of Hatha Yoga in Head and Neck Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sheila Ridner, Martha Rivers Ingram Professor of Nursing, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC SUPP 1282; 1R21CA173202-01 (NIH)
Record Dates: First submitted 2013-09-23; First posted 2013-09-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Head Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Yoga Program for HNC Survivors (Experimental): Following the completion of baseline study measures, participants will be randomized to either do go directly into a Yoga program or to an 8 week wait-list control group. Those in the yoga program will undergo an initial Yoga Evaluation. Patients will receive customized yoga guided practice program, a home practice plan with ongoing modifications. Instructors will assess compliance. A satisfaction assessment is conducted at study-end.
  Interventions: Other: Baseline Study Measures; Behavioral: Yoga Evaluation; Behavioral: Yoga Program; Behavioral: Yoga Practice Plan; Other: Study Assessments
- Wait list control (Active Comparator): Those in the wait list group will have the same assessments as those in the yoga program over the same period of time.
  Interventions: Other: Baseline Study Measures; Other: Study Assessments

INTERVENTIONS:
Other: Baseline Study Measures — Participants will undergo baseline objective and self-report study measures including: 1) ROM in the jaw, neck, and shoulders; 2) posture assessment; 3) pain, and 4) psychological distress. The study measures will take 30-45 minutes to administer.
Behavioral: Yoga Evaluation — The evaluation includes an assessment of nine traditional Yoga components: energy, symptoms, emotions, posture, breathing patterns, gait, muscle/tissue quality, joint flexibility, and muscle strength. Emphasis will be placed on the assessment of jaw/neck/shoulder MSI requiring Yoga practice modification of those poses that are unsafe or not feasible for a patient to perform. Information from the evaluation will be used to establish the tailored Yoga program
  Arms: Modified Yoga Program for HNC Survivors
Behavioral: Yoga Program — The Yoga program has 5 components: 1) Awareness Practice to enhance self-awareness, 2)Poses - 16 core poses will be modified for each patient's specific needs, 3)Breath Work - breath awareness and proper breathing for maximum benefit, 4)Relaxation - alternating between methods of relaxation, 5)Mediation - awareness and practice of inner silence
  Arms: Modified Yoga Program for HNC Survivors
Behavioral: Yoga Practice Plan — To enhance fidelity, a standardized Yoga intervention was chosen that includes postures, meditation, relaxation, and breath work. To ensure safety, the practice plan for each patient will be reviewed prior to initiation. All MSI limitations will be discussed, and appropriate adaptive techniques will be formulated. Qualitative techniques will be used to describe and categorize the types of impairment and modifications. By developing a catalog of impairments and suitable modifications, a safe and uniform Yoga program can be further tested and widely disseminated.
  Arms: Modified Yoga Program for HNC Survivors
Other: Study Assessments — Data collection methods used to assess efficacy include physical measurement/examination, jaw range of motion (device) - scales to measure opening, cervical range of motion(Device), Shoulder Range of Motion - Goniometer, Posture - Wall Zone Grid, self-reported surveys for physical symptoms, pain, psychological symptoms, anxiety, depression and quality of life

SUMMARY:
Treatment for head and neck cancer can result in marked musculo-skeletal impairment (MSI). This study will examine the effects of Hatha Yoga as a therapeutic modality to address MSI.

DETAILED DESCRIPTION:
The use of aggressive treatment for head and neck cancer (HNC) particularly combined modality treatment regimens has resulted in an increase in survival. Unfortunately, this improvement has come with a marked increase in acute and late-effects. Acute HNC treatment-related toxicities have been clearly and extensively documented; however, data pertaining to adverse late-effects, those most likely to impact the survivor's long term symptom burden, functionality, and overall quality of life (QOL), are limited. This pilot study will be conducted to examine the feasibility of tailored Hatha Yoga as a therapeutic modality to address MSI in patients who have survived HNC.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years of age
* >3 months post-treatment of HNC
* no active cancer
* ability to understand English in order to complete questionnaires
* willing to participate in the guided and home Yoga practice
* willing to drive to the study site
* willing and able to provide informed consent
* completed medically indicated physical therapy
* medical clearance by study medical oncologist

Exclusion Criteria:

* a prior cancer diagnosis within the past three years (except basal cell, surgically treated squamous cell skin cancer, early prostate cancer under observation)
* have received radiation therapy or chemotherapy for any condition other than primary HNC
* medical conditions that would prohibit the safe implementation of a Yoga practice (e.g., vertigo, dementia)
* active Yoga practice within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of patients who complete a modified Yoga program for HNC survivors | at 8 weeks
  Number of patients that complete an 8-week course of guided yoga sessions and that complete a Participant Practice Log to document their non-guided home yoga sessions

SECONDARY OUTCOMES:
Change in range of motion (ROM) jaw maximal inter-incisoral opening | at 8 weeks
  Change in ROM from baseline in the jaw maximal inter-incisoral opening, measured in millimeters (mm)
Change in cervical ROM | at 8 weeks
  Change from baseline in cervical ROM, measured in degrees of neck movement
Change in head and neck-related treatment systems | at 8 weeks
  Change from baseline in the Vanderbilt Head and Neck Symptom Survey: 9 questions on treatment-related symptoms with 0 = least amount of problems to 10 = most amount of problems. Higher scores indicate increased treatment-related distress
Change in Brief Pain Inventory | at 8 weeks
  Change from baseline in scores for the Brief Pain Inventory: 9 items with 0 = no pain to 10 = pain as bad as you can imagine. Higher sum of scores indicate greater pain burden
Change in Body Image Quality of Life Inventory | at 8 weeks
  Change from baseline in scores in the Change in Body Image Quality of Life Inventory. 18 questions with minus 3 = very negative effect to plus 3 = very positive effect. sum of scores with higher scores indicating a more positive body image
Change in Anxiety and Depression Scale | 8 weeks
  Change from baseline in scores on the Hospital Anxiety and Depression Inventory with a score of >/= 8 as possible cause for mental health referral

CONTACTS AND LOCATIONS:
Overall Officials: Sheila H Ridner, PhD, RN, Principal Investigator — Vanderbilt University School of Nursing; Barbara Murphy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt University School of Nursing, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/